CLINICAL TRIAL: NCT07344506
Title: Evaluating the Effectiveness of Anti- Ulcerants (Dexlansoprazole, Lansoprazole, and Vonoprazan) With Levofloxacin-based Triple Therapy for Helicobacter Pylori Eradication - A Three-arm Randomized Controlled Trial
Brief Title: CURE-H. Pylori: A Trial on the Combination of Anti-Ulcerants and Levofloxacin-Based Therapy for Helicobacter Pylori Eradication
Acronym: CURE-H Pylori
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-3887
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: H. Pylori Gastrointestinal Disease; H.Pylori Infection; H.Pylori Eradication Rate
Keywords: Helicobacter pylori, Peptic ulcer disease, Combination Triple regime, Dexlansoprazole, Lansoprazole, Vonoprazan, Eradication therapy, Treatment Efficacy; Randomized Controlled Trial; Three Arm
MeSH Terms: conditions — Peptic Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 1: Dexlansoprazole + Levofloxacin-Based Triple Therapy (Experimental): Dexlansoprazole 60mg BD + Levofloxacin 500mg OD + Amoxicillin 1g BD (for 14 days)
  Interventions: Drug: Arm 1: Dexlansoprazole + Levofloxacin-Based Triple Therapy
- Arm 2: Lansoprazole + Levofloxacin-Based Triple Therapy (Experimental): Lansoprazole 30mg BD + Levofloxacin 500mg OD + Amoxicillin 1g BD (for 14 days)
  Interventions: Drug: Arm 2: Lansoprazole + Levofloxacin-Based Triple Therapy
- Arm 3: Vonoprazan + Levofloxacin-Based Triple Therapy (Experimental): Vonoprazan 20mg BD + Levofloxacin 500mg OD + Amoxicillin 1g BD (for 14 days)
  Interventions: Drug: Arm 3: Vonoprazan + Levofloxacin-Based Triple Therapy

INTERVENTIONS:
Drug: Arm 1: Dexlansoprazole + Levofloxacin-Based Triple Therapy — A combination of Dexlansoprazole (60mg twice daily) with Levofloxacin (500mg once daily) and Amoxicillin (1g twice daily) for the eradication of Helicobacter pylori infection.
  Arms: Arm 1: Dexlansoprazole + Levofloxacin-Based Triple Therapy
Drug: Arm 2: Lansoprazole + Levofloxacin-Based Triple Therapy — A combination of Lansoprazole (30mg twice daily) with Levofloxacin (500mg once daily) and Amoxicillin (1g twice daily) for the eradication of Helicobacter pylori infection.
  Arms: Arm 2: Lansoprazole + Levofloxacin-Based Triple Therapy
Drug: Arm 3: Vonoprazan + Levofloxacin-Based Triple Therapy — A combination of Vonoprazan (20mg twice daily) with Levofloxacin (500mg once daily) and Amoxicillin (1g twice daily) for the eradication of Helicobacter pylori infection.
  Arms: Arm 3: Vonoprazan + Levofloxacin-Based Triple Therapy

SUMMARY:
This study, titled CURE-H. Pylori, is a three-arm, parallel-group, open-label, randomized controlled trial designed to evaluate the effectiveness of Dexlansoprazole, Lansoprazole, and Vonoprazan in combination with Levofloxacin and Amoxicillin for Helicobacter pylori eradication. H. pylori infection is a significant health issue worldwide, with an estimated prevalence of 44% globally and around 60% in Pakistan, leading to gastritis, peptic ulcer disease, and increased risks of gastric cancer and mucosa-associated lymphoid tissue lymphoma. Despite the widespread use of PPI-based triple therapies, treatment efficacy has decreased due to increasing antibiotic resistance, especially to Clarithromycin and Metronidazole. This study aims to assess the eradication rate of H. pylori in patients receiving either Dexlansoprazole 60mg, Lansoprazole 30mg, or Vonoprazan 20mg, each combined with Levofloxacin 500mg and Amoxicillin 1g for 14 days. Participants will be randomized into three arms (314 participants per arm) and assessed for H. pylori eradication using a Urea Breath Test (UBT) at follow-up, which will serve as the primary endpoint. Secondary objectives include assessing symptom improvement using the Gastrointestinal Symptom Rating Scale (GSRS), measuring symptoms such as reflux, abdominal pain, indigestion, diarrhea, and constipation. The study will enroll adult patients diagnosed with H. pylori via UBT and who are not currently receiving treatment for the infection. The study will be conducted at healthcare centers in major cities across Pakistan, including Peshawar, Faisalabad, Rawalpindi, Multan, Lahore, Karachi, and Quetta, over a 12-month period. All participants will sign informed consent forms before enrollment, ensuring they understand the study's procedures and risks. Statistical analysis will be performed using SPSS version 26, with categorical variables analyzed using the Chi-square or Fisher's exact test and continuous variables using descriptive statistics. The primary outcome is the H. pylori eradication rate, and secondary outcomes include the improvement in gastrointestinal symptoms. This study is significant because it aims to compare three different PPI-based therapies in the context of H. pylori eradication in a high-resistance population, providing much-needed data for tailoring treatment strategies in regions with high antibiotic resistance like Pakistan. The results could enhance the effectiveness and cost-efficiency of treatment regimens for H. pylori, ultimately improving patient outcomes and reducing the burden of gastric diseases. Ethical approval has been obtained from the Institutional Review Board (IRB) of Dow University of Health Sciences, Karachi, and all procedures will adhere to the principles of human subjects protection. This study will provide valuable insights into the comparative efficacy of different proton pump inhibitors when combined with Levofloxacin-based triple therapy, potentially leading to more effective treatment options for H. pylori infections in Pakistan and similar regions. The total required sample size for this study is 942 participants, with a 20% expected dropout rate. Data collection will be conducted at baseline and six weeks post-treatment, with the aim of addressing the region-specific challenges in H. pylori treatment and contributing to the global knowledge on optimal therapeutic strategies for this infection. Additionally, the trial's findings may contribute to the broader understanding of how regional antibiotic resistance patterns affect treatment outcomes and help shape future guidelines for H. pylori management in endemic areas. This trial will also help assess the safety and tolerability of the different therapies, providing a comprehensive evaluation of both therapeutic efficacy and patient quality of life post-treatment.

DETAILED DESCRIPTION:
Study Title:

CURE-H. Pylori: A Randomized Controlled Trial of Dexlansoprazole, Lansoprazole, and Vonoprazan with Levofloxacin-Based Triple Therapy for Helicobacter pylori Eradication

Study Background:

Helicobacter pylori (H. pylori) infection is a major global health problem, infecting approximately 44% of the population worldwide, with even higher prevalence rates in certain regions. In Pakistan, H. pylori infection affects around 60% of the population, contributing to substantial morbidity and mortality from gastric diseases, including peptic ulcer disease, gastritis, gastric cancer, and mucosa-associated lymphoid tissue lymphoma. The transmission of H. pylori is primarily fecal-oral or oral-oral, often through contaminated water or food, which is exacerbated by poor hygiene and socio-economic conditions. Infection with H. pylori is also a major risk factor for the development of gastric cancer, a leading cause of cancer-related death worldwide.

The standard treatment for H. pylori infection has traditionally been a triple therapy regimen consisting of a proton pump inhibitor (PPI), Amoxicillin, and Clarithromycin. However, the effectiveness of this regimen has decreased significantly in recent years, particularly in areas like Pakistan, where high rates of antibiotic resistance-especially to Clarithromycin and Metronidazole-are prevalent. In addition, many patients are not compliant with prescribed treatments, further decreasing the overall success rates of H. pylori eradication efforts.

Given the importance of effective treatment for H. pylori infection, there is a need for alternative regimens that can overcome resistance to standard antibiotics. Dexlansoprazole, Lansoprazole, and Vonoprazan are all PPIs, but each differs in their pharmacokinetics and mechanism of action. Dexlansoprazole has been shown to have superior pharmacokinetics, with greater maximum plasma concentration and a longer half-life compared to other PPIs. Vonoprazan, a newer PPI, has shown promise in overcoming antibiotic resistance and enhancing the efficacy of antibiotics used in H. pylori eradication. Thus, the combination of these PPIs with Levofloxacin, a broad-spectrum antibiotic, and Amoxicillin may provide an effective alternative to the standard triple therapy, especially in high-resistance regions like Pakistan.

Study Objectives:

The study aims to compare the effectiveness of Dexlansoprazole, Lansoprazole, and Vonoprazan in combination with Levofloxacin and Amoxicillin for the eradication of H. pylori. The specific objectives are:

Primary Objective:

To assess the H. pylori eradication rate in three study groups receiving either Dexlansoprazole, Lansoprazole, or Vonoprazan combined with Levofloxacin-based triple therapy, measured by Urea Breath Test (UBT) at follow-up.

Secondary Objective:

To assess the improvement in gastrointestinal symptoms post-therapy, measured using the Gastrointestinal Symptom Rating Scale (GSRS), which assesses symptoms like reflux, abdominal pain, indigestion, diarrhea, and constipation.

Study Design:

This is a three-arm, parallel-group, open-label, randomized controlled trial (RCT) designed to compare the efficacy of three different PPI-based regimens in the eradication of H. pylori. The study will be conducted over a 12-month period across several healthcare centers in Pakistan, including Peshawar, Faisalabad, Rawalpindi, Multan, Lahore, Karachi, and Quetta. The study aims to recruit a total of 942 participants, with 314 participants per arm, adjusted for a 20% dropout rate.

Methods:

Study Population:

The study will include adult patients (both sexes), diagnosed with H. pylori infection via UBT, who are not currently receiving treatment for H. pylori. Patients must meet the inclusion and exclusion criteria to be eligible for the trial.

Inclusion Criteria:

Adults (≥18 years) of both sexes.

Diagnosed with H. pylori infection through UBT.

Not currently on treatment for H. pylori infection.

Exclusion Criteria:

Pregnant or lactating women.

Patients with severe mental disabilities.

Patients with a history of allergic reactions to any of the drugs used in the study.

Patients who have received antibiotics in the last two weeks before the study.

Randomization:

Participants will be randomly assigned (1:1:1) to one of three treatment arms:

Arm 1: Dexlansoprazole 60mg BD + Levofloxacin 500mg OD + Amoxicillin 1g BD (for 14 days).

Arm 2: Lansoprazole 30mg BD + Levofloxacin 500mg OD + Amoxicillin 1g BD (for 14 days).

Arm 3: Vonoprazan 20mg BD + Levofloxacin 500mg OD + Amoxicillin 1g BD (for 14 days).

Randomization will ensure unbiased allocation of participants to the treatment arms.

Data Collection:

Data will be collected at two points in time:

Baseline: Prior to the initiation of treatment, demographic information, medical history, and baseline symptoms using GSRS will be collected.

Follow-up (6 weeks): At the follow-up visit, participants will undergo the UBT to assess H. pylori eradication, and their gastrointestinal symptoms will be reassessed using GSRS.

A self-reporting questionnaire will gather information on various factors, including the use of NSAIDs, previous antibiotics, alcohol consumption, smoking history, and more.

Outcome Measures:

Primary Outcome:

The H. pylori eradication rate will be measured as the percentage of participants in each arm who have a negative UBT after completing the 14-day treatment regimen.

Secondary Outcomes:

Gastrointestinal Symptom Improvement: Measured by the GSRS, which evaluates symptoms like reflux, abdominal pain, indigestion, diarrhea, and constipation.

Adverse Events: The occurrence of any side effects or adverse events related to the treatments will be monitored throughout the trial.

Statistical Analysis:

Statistical analysis will be performed using SPSS version 26. Descriptive statistics will be used to summarize the baseline characteristics of the participants. The primary outcome (H. pylori eradication rate) will be analyzed using Chi-square or Fisher's exact tests. Continuous variables, such as symptom scores, will be analyzed using t-tests or ANOVA where appropriate. An intention-to-treat analysis will be performed to include all randomized participants, regardless of adherence. A p-value < 0.05 will be considered statistically significant.

Ethical Considerations:

The study has received approval from the Institutional Review Board (IRB) of Dow University of Health Sciences, Karachi. Participants will be fully informed about the study's purpose, procedures, risks, and benefits, and will sign an informed consent form before enrollment. The study will adhere to ethical guidelines for research involving human participants, ensuring confidentiality and voluntary participation.

Study Timeline:

Preparation Phase:

Ethical approval, participant recruitment, and site preparation (1-2 months).

Enrollment Phase:

Recruitment of 942 participants (3-4 months).

Intervention Phase:

Participants will receive the prescribed treatment for 14 days (12 months).

Follow-up Phase:

Data collection at baseline and six weeks post-treatment (12 months).

Expected Impact:

The study aims to provide valuable insights into the most effective PPI-based regimen for H. pylori eradication in regions with high antibiotic resistance, particularly in Pakistan. By comparing Dexlansoprazole, Lansoprazole, and Vonoprazan in combination with Levofloxacin and Amoxicillin, this study could lead to more effective, region-specific treatment regimens, addressing the growing challenge of antibiotic resistance. The findings will contribute to global knowledge of H. pylori treatment and may lead to new, more effective therapeutic strategies for countries with similar antibiotic resistance profiles.

The study's findings could also inform the development of patient-centered treatment plans that take into account regional resistance patterns, leading to improved patient outcomes and reduced healthcare costs. Furthermore, this research will help shape future guidelines for H. pylori management and could lead to the wider adoption of Vonoprazan and Dexlansoprazole in clinical practice.

Conclusion:

This trial will provide crucial data on the comparative effectiveness of PPI-based triple therapies in H. pylori eradication. The results are expected to contribute significantly to the treatment landscape in Pakistan and other regions with similar healthcare challenges. If successful, the study could have wide-reaching implications for gastroenterology and infectious disease management, particularly in addressing the growing issue of antibiotic resistance. The evidence generated could ultimately enhance the quality of life for millions of individuals suffering from H. pylori-related diseases, while also informing public health strategies aimed at reducing the global burden of gastric cancer and other gastrointestinal disorders.

ELIGIBILITY:
Inclusion Criteria:

Adult patients of both sexes, presenting to the out-patient departments of the participating healthcare centres, and diagnosed through a UBT to have H.Pylori infection by their physician will be eligible for enrolment in the study, but are currently not receiving any treatment for H.Pylori infection.

Exclusion Criteria:

1. Those who will not provide written consent for the study.
2. Patients with severe mental disability,
3. pregnant or lactating women,
4. those who are already on treatment for H.Pylori infection, and
5. those who have received any antibiotic within the last two weeks of enrolling in this study will be excluded.
6. Patients with known previous documented drug allergies for the current regime will be excluded from the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 942 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
H. pylori Eradication | 2 years
  The primary outcome is the eradication rate of H. pylori, measured by a negative Urea Breath Test (UBT) after the completion of the 14-day treatment regimen in each of the three arms.
  A successful eradication is defined as a negative UBT performed four weeks after completing the treatment.
  The eradication rate will be compared between the three arms: Dexlansoprazole + Levofloxacin-based triple therapy, Lansoprazole + Levofloxacin-based triple therapy, and Vonoprazan + Levofloxacin-based triple therapy.

SECONDARY OUTCOMES:
Gastrointestinal Symptom Improvement: | 2 years
  The improvement in gastrointestinal symptoms will be measured using the Gastrointestinal Symptom Rating Scale (GSRS), which assesses symptoms related to reflux, abdominal pain, indigestion, diarrhea, and constipation.
  The GSRS will be administered at both baseline (before treatment initiation) and follow-up (six weeks after treatment completion) to assess symptom improvement in each treatment group.
Adverse Events | 2 years
  The occurrence of adverse events related to the treatment regimen (e.g., nausea, diarrhea, abdominal pain, dizziness, headache) will be monitored and reported.
  These events will be recorded to evaluate the safety and tolerability of the three treatment regimens.
Treatment Compliance | 2 years
  Participants will be monitored for treatment adherence, defined as taking at least 80% of the prescribed medication.
  Reasons for non-adherence will be recorded, if applicable.

CONTACTS AND LOCATIONS:
Locations (1):
- Sindh Institute of Advanced Endoscopy and Gastroenterology (SIAG), DUHS, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
The decision about data sharing will be made after study completion, and further details will be available at that time